CLINICAL TRIAL: NCT00652626
Title: A Phase 1, Open-Label, Multi-Center, Parallel Group Study to the Pharmacokinetics and Safety of Subcutaneous Azacitidine in Adult Cancer Patients With and Without Impaired Renal Function
Brief Title: Pharmacokinetics and Safety Study of Azacitidine in Cancer Patients With and Without Impaired Renal Function
Acronym: RENAL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AZA PH US 2007 PK006
Record Dates: First submitted 2008-04-01; First posted 2008-04-04 (Estimated); Results first posted 2013-10-17 (Estimated); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: MDS; AML; Solid Tumors; Multiple Myeloma; Non-Hodgkin's Lymphoma; Hodgkin's Disease
Keywords: MDS; AML; Solid Tumors; Azacitidine; PK; Pharmacokinetics; Renal Impairment; Multiple Myeloma; Non-Hodgkin's Lymphoma; Hodgkin's Disease
MeSH Terms: conditions — Multiple Myeloma; Lymphoma, Non-Hodgkin; Hodgkin Disease; Renal Insufficiency | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Azacitidine 25 mg/m^2 (Experimental): Participants with normal renal function received a single subcutaneous dose of azacitidine 25 mg/m^2 on Day 1. Participants could continue treatment in the extension phase, which allowed up to 6 cycles of treatment with 75 mg/m^2 daily on Days 1-7 of each 28-day cycle.
  Interventions: Drug: azacitidine
- Azacitidine 50 mg/m^2 (Experimental): Participants with normal renal function received a single subcutaneous dose of azacitidine 50 mg/m^2 on Day 1. Participants could continue treatment in the extension phase, which allowed up to 6 cycles of treatment with 75 mg/m^2 daily on Days 1-7 of each 28-day cycle.
  Interventions: Drug: azacitidine
- Azacitidine 75 mg/m^2 (Experimental): Participants with normal renal function received subcutaneous doses of azacitidine 75 mg/m^2 on Days 1 to 5. Participants could continue treatment in the extension phase, which allowed up to 6 cycles of treatment with 75 mg/m^2 daily on Days 1-7 of each 28-day cycle.
  Interventions: Drug: azacitidine
- Azacitidine 100 mg/m^2 (Experimental): Participants with normal renal function received a single subcutaneous dose of azacitidine 100 mg/m^2 on Day 1. Participants could continue treatment in the extension phase, which allowed up to 6 cycles of treatment with 75 mg/m^2 daily on Days 1-7 of each 28-day cycle.
  Interventions: Drug: azacitidine
- Severe RI: azacitidine 75 mg/m^2 (Experimental): Participants with severe renal impairment (RI; defined as creatinine clearance < 30 mL/min/1.73 m^2) received subcutaneous doses of azacitidine 75 mg/m^2 on Days 1 to 5. Participants could continue treatment in the extension phase, which allowed up to 6 cycles of treatment with 75 mg/m^2 daily on Days 1-7 of each 28-day cycle.
  Interventions: Drug: azacitidine

INTERVENTIONS:
Drug: azacitidine
  Other Names: Vidaza

SUMMARY:
The purpose of this study is to evaluate three things. The first being whether azacitidine is absorbed in the body at the same rate or proportion for different concentrations. The second is to determine the effect renal impairment has or does not have on the absorption of azacitidine. The third is to determine if azacitidine is safe and well tolerated in patients with renal function impairment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of one of the following:

  * MDS according to the French-American-British (FAB) classification system: refractory anemia (RA), refractory anemia with ringed sideroblasts (RARS), refractory anemia with excess blasts (RAEB), refractory anemia with excess blasts in transformation (RAEB-T), or chronic myelomonocytic leukemia (CMML); or
  * Acute myelogenous leukemia (AML) in remission,
  * Malignant solid tumor,
  * Multiple myeloma (MM),
  * Non-Hodgkin lymphoma (NHL), or
  * Hodgkin lymphoma (HD)
* Patients with a history of treated brain metastases should be clinically stable for greater than 4 weeks prior to signing the informed consent form and off glucocorticoid therapy for central nervous system (CNS) edema for at least 4 weeks
* Be capable of giving informed consent
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Have a life expectancy ≥ 3 months
* Have stable renal function for at least 2 months
* Have average calculated creatinine clearance of:

  * >80 mL/min/1.73m^2 for Cohorts 1, 2, 3, and 4
  * <30 mL/min/1.73m^2 for Cohort 5 - Severe renal impairment,
  * 50-80 mL/min/1.73m^2 for Cohort 6 - Mild renal impairment,
  * 30 to <50 mL/min/1.73m^2 for Cohort 7 - Moderate renal impairment
* Have organ and marrow function at the screening and pre-dose visits as defined below:

  * Hemoglobin ≥8 g/dL,
  * Absolute neutrophil count ≥0.75 x 10^3/µL,
  * Platelets ≥30 x 10^3/µL,
  * Total bilirubin ≤1.5 times the upper limit of normal (ULN),
  * Aspartate aminotransferase (AST) ≤2 times the ULN, and
  * Alanine transaminase (ALT) ≤2 times the ULN;
* Have a 12-lead electrocardiogram (ECG) that is not clinically significant, as determined by the Investigator, at screening
* Have serum bicarbonate:

  * 20 mEq/L for patients with normal renal function (cohorts 1, 2, 3 and 4),
  * 16 mEq/L for patients with impaired renal function (cohorts 5, 6 and 7)
* Women of childbearing potential may participate, providing are not pregnant and agree to use at least 2 effective contraceptive methods throughout the study
* Males with a female partner of childbearing potential must agree to use at least 2 effective contraceptive methods throughout the study and to avoid fathering a child for 6 months following the date of the last dose of study medication
* Be a nonsmoker or must not have smoked for at least 30 days before the screening visit and agree to abstain from smoking during study participation

Exclusion Criteria:

* Women who are pregnant or nursing;
* Had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to signing informed consent
* Have been treated with an investigational agent within 4 weeks prior to signing the informed consent form
* Have ongoing clinically significant adverse event(s) due to chemotherapy, radiotherapy or investigational agents administered more than 4 weeks prior to signing the informed consent as determined by the Investigator
* Have known or suspected hypersensitivity to azacitidine or mannitol
* Have an uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia
* Have low blood pressure (supine blood pressure <90/60 mmHg)
* Have human immunodeficiency virus (HIV), or active hepatitis virus B or C
* Have advanced malignant hepatic tumors
* Have end stage renal disease requiring dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2008-11-01 (Actual); Primary Completion 2012-07-01 (Actual); Study Completion 2012-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay Backstrom, MD, Study Director — Celgene Corporation
Locations (11):
- United States (11):
  - Sutter East Bay Hospitals, Berkeley, California
  - Palm Springs Research Institute, Hialeah, Florida
  - MCG Cancer Center, Augusta, Georgia
  - Joliet Oncology-Hematology Associates, Ltd., Joliet, Illinois
  - University of Kentucky-Markey Cancer Center Clinical Research Organization, Lexington, Kentucky
  - Nevada Cancer Institute, Las Vegas, Nevada
  - Montefiore Medical Center, The Bronx, New York
  - Mid Dakota Clinical P.C. - Cancer Treatment and Research Center, Bismarck, North Dakota
  - Gabrail Cancer Center, Canton, Ohio
  - Pharma Resource, East Providence, Rhode Island
  - Cancer Therapy and Research Center, San Antonio, Texas

REFERENCES:
- [Background] Wehmeyer J, Zaiss M, Losem C, Schmitz S, Niemeier B, Harde J, Hannig CV, Harich HD, Muller J, Klausmann M, Tessen HW, Potthoff K. Impact of performance status and transfusion dependency on outcome of patients with myelodysplastic syndrome, acute myeloid leukemia and chronic myelomonocytic leukemia treated with azacitidine (PIAZA study). Eur J Haematol. 2018 Dec;101(6):766-773. doi: 10.1111/ejh.13160. Epub 2018 Oct 25. PMID 30091166
- [Background] Platzbecker U, Middeke JM, Sockel K, Herbst R, Wolf D, Baldus CD, Oelschlagel U, Mutherig A, Fransecky L, Noppeney R, Bug G, Gotze KS, Kramer A, Bochtler T, Stelljes M, Groth C, Schubert A, Mende M, Stolzel F, Borkmann C, Kubasch AS, von Bonin M, Serve H, Hanel M, Duhrsen U, Schetelig J, Rollig C, Kramer M, Ehninger G, Bornhauser M, Thiede C. Measurable residual disease-guided treatment with azacitidine to prevent haematological relapse in patients with myelodysplastic syndrome and acute myeloid leukaemia (RELAZA2): an open-label, multicentre, phase 2 trial. Lancet Oncol. 2018 Dec;19(12):1668-1679. doi: 10.1016/S1470-2045(18)30580-1. Epub 2018 Nov 12. PMID 30442503
- [Background] Stevens B, Winters A, Gutman JA, Fullerton A, Hemenway G, Schatz D, Miltgen N, Wei Q, Abbasi T, Vali S, Singh NK, Drusbosky L, Cogle CR, Hammes A, Abbott D, Jordan CT, Smith C, Pollyea DA. Sequential azacitidine and lenalidomide for patients with relapsed and refractory acute myeloid leukemia: Clinical results and predictive modeling using computational analysis. Leuk Res. 2019 Jun;81:43-49. doi: 10.1016/j.leukres.2019.04.005. Epub 2019 Apr 13. PMID 31009835
- [Background] Laille E, et al. A 2-Part Phase I Study in Patients with Solid or Hematologic Malignancies: Dose Proportionality of Subcutaneous (SC) Azacitidine (AZA) and Pharmacokinetics of SC AZA in Patients with Severe Renal Impairment . Presented at American Society of Hematology 2011, December 10-13, 2011, San Diego, CA. Abstract No. 3480.
- [Background] Du X, Lai YY, Xiao Z, Liu T, Hu Y, Sun A, Li X, Shen ZX, Jin J, Yu L, Laille E, Dong Q, Songer S, Beach CL. Efficacy, safety and pharmacokinetics of subcutaneous azacitidine in Chinese patients with higher risk myelodysplastic syndromes: Results from a multicenter, single-arm, open-label phase 2 study. Asia Pac J Clin Oncol. 2018 Jun;14(3):270-278. doi: 10.1111/ajco.12835. Epub 2017 Dec 28. PMID 29282890

RESULTS

PARTICIPANT FLOW:
Groups:
- Azacitidine 25 mg/m^2: Participants with normal renal function (defined as creatinine clearance > 80 mL/min/1.73m^2) received a single subcutaneous dose of azacitidine 25 mg/m^2 on Day 1.
- Azacitidine 50 mg/m^2: Participants with normal renal function received a single subcutaneous dose of azacitidine 50 mg/m^2 on Day 1.
- Azacitidine 75 mg/m^2: Participants with normal renal function received subcutaneous doses of azacitidine 75 mg/m^2 on Days 1 to 5.
- Azacitidine 100 mg/m^2: Participants with normal renal function received a single subcutaneous dose of azacitidine 100 mg/m^2 on Day 1.
- Severe RI: Azacitidine 75 mg/m^2: Participants with severe renal impairment (RI; defined as creatinine clearance < 30 mL/min/1.73 m^2) received subcutaneous doses of azacitidine 75 mg/m^2 on Days 1 to 5.
- Extension Phase: Normal RF: Participants with normal renal function (RF) received up to 6 cycles of treatment with 75 mg/m^2 azacitidine daily on Days 1-7 of each 28-day cycle.
- Extension Phase: Severe RI: Participants with severe renal impairment (RI) received up to 6 cycles of treatment with 75 mg/m^2 azacitidine daily on Days 1-7 of each 28-day cycle.
Period: Initial Treatment Phase
Arm/Group | Azacitidine 25 mg/m^2 | Azacitidine 50 mg/m^2 | Azacitidine 75 mg/m^2 | Azacitidine 100 mg/m^2 | Severe RI: Azacitidine 75 mg/m^2 | Extension Phase: Normal RF | Extension Phase: Severe RI
Started | 5 | 5 | 7 | 6 | 8 | 0 | 0
Received Study Drug | 5 | 5 | 6 | 5 | 6 | 0 | 0
Completed | 5 | 5 | 6 | 5 | 5 | 0 | 0
Not Completed | 0 | 0 | 1 | 1 | 3 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Sponsor Request | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0 | 0
Period: Extension Phase
Arm/Group | Azacitidine 25 mg/m^2 | Azacitidine 50 mg/m^2 | Azacitidine 75 mg/m^2 | Azacitidine 100 mg/m^2 | Severe RI: Azacitidine 75 mg/m^2 | Extension Phase: Normal RF | Extension Phase: Severe RI
Started | 0 | 0 | 0 | 0 | 0 | 14 | 4
Completed | 0 | 0 | 0 | 0 | 0 | 2 (A participant was considered completed if they had completed 6 cycles of therapy.) | 1 (A participant was considered completed if they had completed 6 cycles of therapy.)
Not Completed | 0 | 0 | 0 | 0 | 0 | 12 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 2 | 1
Not completed — No Longer Receiving Clinical Benefit | 0 | 0 | 0 | 0 | 0 | 6 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety population. The total number of participants in the study was 27; 18 continued treatment in the extension phase.
Groups:
- Total: Total of all reporting groups
Arm/Group | Azacitidine 25 mg/m^2 | Azacitidine 50 mg/m^2 | Azacitidine 75 mg/m^2 | Azacitidine 100 mg/m^2 | Severe RI: Azacitidine 75 mg/m^2 | Extension Phase: Normal RF | Extension Phase: Severe RI | Total
Number analyzed (Participants) | 5 | 5 | 6 | 5 | 6 | 14 | 4 | 45
Age, Continuous [Mean (Standard Deviation); unit: years]
  Initial Treatment Period | 67.6 (3.78) | 64.6 (9.63) | 53.5 (10.19) | 57.0 (12.02) | 74.5 (12.58) | NA (NA) — Data for provided initial treatment period arms only | NA (NA) — Data provided for initial treatment period arms only | 63.5 (12.32)
  Extension Treatment Period | NA (NA) — Data provided for extension treatment period arms only | NA (NA) — Data provided for extension treatment period arms only | NA (NA) — Data provided for extension treatment period arms only | NA (NA) — Data provided for extension treatment period arms only | NA (NA) — Data provided for extension treatment period arms only | 60.6 (9.52) | 68.8 (11.0) | 62.4 (10.15)
Sex/Gender, Customized [Number; unit: participants] — Data provided for initial treatment phase groups only.
  participants
    Female | 3 | 3 | 3 | 4 | 3 | 0 | 0 | 16
    Male | 2 | 2 | 3 | 1 | 3 | 0 | 0 | 11
Race/Ethnicity, Customized [Number; unit: participants] — Data provided for initial treatment phase groups only.
  participants
    Black | 1 | 2 | 1 | 2 | 2 | 0 | 0 | 8
    White | 4 | 3 | 5 | 3 | 4 | 0 | 0 | 19
Region of Enrollment [Number; unit: participants] — Data provided for initial treatment phase groups only.
  participants
    United States | 5 | 5 | 6 | 5 | 6 | 0 | 0 | 27
Gender of Extension Period Participants [Number; unit: participants]
  Female | 0 | 0 | 0 | 0 | 0 | 8 | 2 | 10
  Male | 0 | 0 | 0 | 0 | 0 | 6 | 2 | 8
Race: Extension Phase [Number; unit: participants]
  Black | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 5
  White | 0 | 0 | 0 | 0 | 0 | 9 | 4 | 13
Eastern Cooperative Oncology Group (ECOG) Performance Status: Initial Treatment Phase [Number; unit: participants] — Scale used by doctors and researchers to assess how a patient's disease is progressing, assess how the disease affects the daily living abilities of the patient, and determine appropriate treatment and prognosis. 0 = fully active, no restrictions; 1 = restricted but ambulatory and capable of light work; 2 = ambulatory and capable of self-care but unable to work. 3 = Capable of only limited self care, confined to bed or chair more than 50% of waking hours. 4 = Completely disabled. Cannot carry on any self care. Totally confined to bed or chair. 5 = Dead.
  participants
    0 | 2 | 2 | 1 | 0 | 2 | 0 | 0 | 7
    1 | 3 | 3 | 4 | 5 | 3 | 0 | 0 | 18
    2 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2
Eastern Cooperative Oncology Group (ECOG) Performance Status: Extension Phase [Number; unit: participants]
  0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 3
  1 | 0 | 0 | 0 | 0 | 0 | 11 | 3 | 14
  2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Body Surface Area (BSA) [Mean (Standard Deviation); unit: m^2]
  Initial Treatment Period | 2.0 (0.20) | 1.9 (0.28) | 1.9 (0.42) | 1.6 (0.15) | 1.8 (0.15) | NA (NA) — Data provided for initial treatment period arms only | NA (NA) — Data provided for initial treatment period arms only | 1.9 (0.27)
  Extension Period | NA (NA) — Data provided for extension treatment period arms only | NA (NA) — Data provided for extension treatment period arms only | NA (NA) — Data provided for extension treatment period arms only | NA (NA) — Data provided for extension treatment period arms only | NA (NA) — Data provided for extension treatment period arms only | 1.9 (0.35) | 1.9 (0.06) | 1.9 (0.31)
Cancer Diagnosis: Initial Treatment Phase [Number; unit: participants] — MDS = myelodysplastic syndrome; MM = multiple myeloma; RA = refractory anemia; RAEB-T = refractory anemia with excess blasts in transformation; RARS = refractory anemia with ringed sideroblasts; CMML = chronic myelomonocytic leukemia.
  participants
    Myelodysplastic syndrome-RA | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2
    Myelodysplastic syndrome-RARS | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
    Myelodysplastic syndrome-RAEB-T | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2
    Chronic myelomonocytic leukemia | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
    Solid tumor | 3 | 3 | 5 | 5 | 4 | 0 | 0 | 20
    Multiple myeloma | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cancer Diagnosis: Extension Phase [Number; unit: participants]
  Myelodysplastic syndrome-RA | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Myelodysplastic syndrome-RARS | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Myelodysplastic syndrome-RAEB-T | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Chronic myelomonocytic leukemia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Solid tumor | 0 | 0 | 0 | 0 | 0 | 12 | 3 | 15
  Multiple myeloma | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to 8 Hours Post-dose
Description: Area under the plasma concentration-time curve from time 0 to 8 hours post-dose (AUC0-8) of azacitidine following a single dose of azacitidine on Day 1, calculated by the linear trapezoidal rule.
Time Frame: Day 1 at predose, 5, 15, 30, 45 minutes and 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, and 8 hours post-dose
Population: Pharmacokinetic (PK) Population, consisting of all participants with evaluable plasma or urine concentration data for azacitidine. This analysis was performed for participants with normal renal function only.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Azacitidine 25 mg/m^2 | Azacitidine 50 mg/m^2 | Azacitidine 75 mg/m^2 | Azacitidine 100 mg/m^2
Number analyzed (Participants) | 5 | 5 | 6 | 5
ng*hr/mL | 455.86 (26.04) | 897.43 (31.00) | 921.87 (39.215) | 1502.86 (25.57)

2. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the Last Quantifiable Time Point
Description: Area under the plasma concentration-time curve from time zero to the last quantifiable time point (AUC0-t) of azacitidine following a single dose of azacitidine on Day 1, calculated by the linear trapezoidal rule.
Time Frame: Day 1 at predose, 5, 15, 30, 45 minutes and 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, and 8 hours post-dose
Population: Pharmacokinetic Population, consisting of all participants with evaluable plasma or urine concentration data for azacitidine. This analysis was performed for participants with normal renal function only.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Azacitidine 25 mg/m^2 | Azacitidine 50 mg/m^2 | Azacitidine 75 mg/m^2 | Azacitidine 100 mg/m^2
Number analyzed (Participants) | 5 | 5 | 6 | 5
ng*hr/mL | 454.80 (26.22) | 895.38 (31.20) | 920.76 (39.20) | 1505.16 (25.57)
Statistical Analysis 1: Comparison: Azacitidine 25 mg/m^2 vs Azacitidine 50 mg/m^2; Geometric means, ratio and 90% confidence interval (CI) of ratio of geometric means are from one way analysis of variance models on the nature log-transformed dose-normalized AUC0-t, obtained on Day 1. Azacitidine 25 mg/m^2 is the reference group for comparisons; Test type: Superiority or Other; Ratio (%) of Geometric Means = 98.4, 90% CI 2-sided [64.0 to 151.3] — Ratio of geometric means is calculated as Azacitidine 50 mg/m^2 / Azacitidine 25 mg/m^2 and expressed as a percentage
Statistical Analysis 2: Comparison: Azacitidine 25 mg/m^2 vs Azacitidine 75 mg/m^2; Geometric means, ratio and 90% CI of ratio of geometric means are from one way analysis of variance models on the nature log-transformed dose-normalized AUC0-t, obtained on Day 1. Azacitidine 25 mg/m^2 is the reference group for comparisons; Test type: Superiority or Other; Ratio (%) of Geometric Means = 67.5, 90% CI 2-sided [44.7 to 101.8] — Ratio of geometric means is calculated as Azacitidine 75 mg/m^2 / Azacitidine 25 mg/m^2 and expressed as a percentage
Statistical Analysis 3: Comparison: Azacitidine 25 mg/m^2 vs Azacitidine 100 mg/m^2; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; Ratio (%) of Geometric Means = 82.7, 90% CI 2-sided [53.8 to 127.2] — Ratio of geometric means is calculated as Azacitidine 100 mg/m^2 / Azacitidine 25 mg/m^2 and expressed as a percentage

3. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Infinity
Description: The area under the plasma concentration-time curve from time zero to infinity (AUC0-inf) for azacitidine after a single dose, calculated by the linear trapezoidal rule and extrapolated to infinity according to the following equation:
  AUC0-inf = AUC0-t + (Ct/ke), where Ct is the last quantifiable concentration and ke = elimination rate constant.
Time Frame: Day 1 at predose, 5, 15, 30, 45 minutes and 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, and 8 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Azacitidine 25 mg/m^2 | Azacitidine 50 mg/m^2 | Azacitidine 75 mg/m^2 | Azacitidine 100 mg/m^2
Number analyzed (Participants) | 5 | 5 | 6 | 5
ng*hr/mL | 460.47 (25.79) | 897.42 (30.93) | 945.50 (39.05) | 1533.37 (23.96)
Statistical Analysis 1: Comparison: Azacitidine 25 mg/m^2 vs Azacitidine 50 mg/m^2; Geometric means, ratio and 90% CI of ratio of geometric means are from one way analysis of variance models on the nature log-transformed dose-normalized AUC0-inf, obtained on Day 1. Azacitidine 25 mg/m^2 is the reference group for comparisons; Test type: Superiority or Other; Ratio (%) of Geometric Means = 97.4, 90% CI 2-sided [63.8 to 148.8] — Ratio of geometric mean is calculated as Azacitidine 50 mg/m^2 / Azacitidine 25 mg/m^2 and expressed as a percentage
Statistical Analysis 2: Comparison: Azacitidine 25 mg/m^2 vs Azacitidine 75 mg/m^2; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; Ratio (%) of Geometric Means = 68.5, 90% CI 2-sided [45.7 to 102.7] — Ratio of geometric mean is calculated as Azacitidine 75 mg/m^2 / Azacitidine 25 mg/m^2 and expressed as a percentage
Statistical Analysis 3: Comparison: Azacitidine 25 mg/m^2 vs Azacitidine 100 mg/m^2; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; Ratio (%) of Geometric Means = 83.2, 90% CI 2-sided [54.5 to 127.1] — Ratio of geometric mean is calculated as Azacitidine 100 mg/m^2 / Azacitidine 25 mg/m^2 and expressed as a percentage

4. Primary Outcome: Maximum Plasma Concentration of Azacitidine (Cmax)
Description: The maximum observed plasma concentration of azacitidine after a single dose on Day 1.
Time Frame: Day 1 at predose, 5, 15, 30, 45 minutes and 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, and 8 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Azacitidine 25 mg/m^2 | Azacitidine 50 mg/m^2 | Azacitidine 75 mg/m^2 | Azacitidine 100 mg/m^2
Number analyzed (Participants) | 5 | 5 | 6 | 5
ng/mL | 293.38 (34.11) | 749.04 (61.03) | 745.50 (57.90) | 1261.96 (39.19)
Statistical Analysis 1: Comparison: Azacitidine 25 mg/m^2 vs Azacitidine 50 mg/m^2; Geometric means, ratio and 90% CI of ratio of geometric means are from one way analysis of variance models on the nature log-transformed dose-normalized Cmax, obtained on Day 1. Azacitidine 25 mg/m^2 is the reference group for comparisons; Test type: Superiority or Other; Ratio (%) of Geometric Means = 127.7, 90% CI 2-sided [66.3 to 245.7] — Ratio of geometric means is calculated as Azacitidine 50 mg/m^2 / Azacitidine 25 mg/m^2 and expressed as a percentage
Statistical Analysis 2: Comparison: Azacitidine 25 mg/m^2 vs Azacitidine 75 mg/m^2; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; Ratio (%) of Geometric Means = 84.7, 90% CI 2-sided [45.3 to 158.5] — Ratio of geometric means is calculated as Azacitidine 75 mg/m^2 / Azacitidine 25 mg/m^2 and expressed as a percentage
Statistical Analysis 3: Comparison: Azacitidine 25 mg/m^2 vs Azacitidine 100 mg/m^2; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; Ratio (%) of Geometric Means = 107.5, 90% CI 2-sided [55.9 to 207.0] — Ratio of geometric means is calculated as Azacitidine 100 mg/m^2 / Azacitidine 25 mg/m^2 and expressed as a percentage

5. Primary Outcome: Time to Maximum Plasma Concentration of Azacitidine (Tmax)
Description: The time to first maximum observed plasma concentration of azacitidine after a single dose on Day 1.
Time Frame: Day 1 at predose, 5, 15, 30, 45 minutes and 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, and 8 hours post-dose
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Azacitidine 25 mg/m^2 | Azacitidine 50 mg/m^2 | Azacitidine 75 mg/m^2 | Azacitidine 100 mg/m^2
Number analyzed (Participants) | 5 | 5 | 6 | 5
hours | 0.25 [0.25 to 1.00] | 0.25 [0.25 to 0.78] | 0.25 [0.25 to 0.50] | 0.27 [0.25 to 0.75]

6. Primary Outcome: Terminal Phase Half-life of Azacitidine (t½)
Description: The terminal phase half-life of azacitidine after a single dose on Day 1, calculated according to the following equation: t½ = 0.693/λz, where λz is the terminal phase rate constant.
Time Frame: Day 1 at predose, 5, 15, 30, 45 minutes and 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, and 8 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Azacitidine 25 mg/m^2 | Azacitidine 50 mg/m^2 | Azacitidine 75 mg/m^2 | Azacitidine 100 mg/m^2
Number analyzed (Participants) | 5 | 5 | 6 | 5
hours | 1.38 (27.31) | 0.63 (35.72) | 1.19 (102.56) | 1.03 (78.48)

7. Primary Outcome: Apparent Total Clearance of Azacitidine (CL/F)
Description: The apparent total clearance of azacitidine after a single dose on Day 1, calculated as Dose/AUC0-inf.
Time Frame: Day 1 at predose, 5, 15, 30, 45 minutes and 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, and 8 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters/hour
Arm/Group | Azacitidine 25 mg/m^2 | Azacitidine 50 mg/m^2 | Azacitidine 75 mg/m^2 | Azacitidine 100 mg/m^2
Number analyzed (Participants) | 5 | 5 | 6 | 5
liters/hour | 104.58 (25.00) | 105.76 (17.03) | 151.55 (30.88) | 106.00 (25.64)
Statistical Analysis 1: Comparison: Azacitidine 25 mg/m^2 vs Azacitidine 50 mg/m^2; Geometric means, ratio and 90% CI of ratio of geometric means are from one way analysis of variance model on the nature log-transformed CL/F obtained on Day 1. Azacitidine 25 mg/m^2 is the reference group for comparisons; Test type: Superiority or Other; Ratio (%) of Geometric Means = 101.1, 90% CI 2-sided [71.2 to 143.6] — Ratio of geometric mean is calculated as Azacitidine 50 mg/m^2 / Azacitidine 25 mg/m^2 and expressed as a percentage
Statistical Analysis 2: Comparison: Azacitidine 25 mg/m^2 vs Azacitidine 75 mg/m^2; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; Ratio (%) of Geometric Means = 144.9, 90% CI 2-sided [103.6 to 202.7] — Ratio of geometric mean is calculated as Azacitidine 75 mg/m^2 / Azacitidine 25 mg/m^2 and expressed as a percentage
Statistical Analysis 3: Comparison: Azacitidine 25 mg/m^2 vs Azacitidine 100 mg/m^2; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; Ratio (%) of Geometric Means = 101.4, 90% CI 2-sided [71.4 to 143.9] — Ratio of geometric mean is calculated as Azacitidine 100 mg/m^2 / Azacitidine 25 mg/m^2 and expressed as a percentage

8. Primary Outcome: Apparent Volume of Distribution of Azacitidine (Vz/F)
Description: The apparent volume of distribution of azacitidine after a single dose on Day 1, calculated according to the equation: Vz/F = Apparent total clearance (CL/F) / terminal phase rate constant (λz)
Time Frame: Day 1 at predose, 5, 15, 30, 45 minutes and 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, and 8 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Azacitidine 25 mg/m^2 | Azacitidine 50 mg/m^2 | Azacitidine 75 mg/m^2 | Azacitidine 100 mg/m^2
Number analyzed (Participants) | 5 | 5 | 6 | 5
liters | 208.69 (45.57) | 96.74 (36.75) | 259.44 (121.71) | 456.69 (99.41)

9. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to 8 Hours Post-dose After Single and Multiple Doses of Azacitidine
Description: The effect of renal impairment on azacitidine pharmacokinetics was analyzed by comparing PK parameters obtained on Days 1 and 5 from participants with severe renal impairment and those with normal renal function.
  Area under the plasma concentration-time curve from time 0 to 8 hours post-dose (AUC0-8) of azacitidine following a single dose (Day 1) and multiple doses (Day 5) was calculated by the linear trapezoidal rule.
Time Frame: Day 1 and Day 5: predose, 5, 15, 30, 45 minutes and 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, and 8 hours post-dose
Population: Pharmacokinetic Population, consisting of all participants with evaluable plasma or urine concentration data for azacitidine. This analysis was performed for participants in the 2 treatment groups who received azacitidine treatment for 5 days.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Groups:
- Normal RF: Azacitidine 75 mg/m^2: Participants with normal renal function (RF) received subcutaneous doses of azacitidine 75 mg/m^2 on Days 1 to 5.
- Severe RI: Azacitidine 75 mg/m^2: Participants with severe renal impairment (RI) received subcutaneous doses of azacitidine 75 mg/m^2 on Days 1 to 5.
Arm/Group | Normal RF: Azacitidine 75 mg/m^2 | Severe RI: Azacitidine 75 mg/m^2
Number analyzed (Participants) | 6 | 6
ng*hr/mL
  Day 1 | 921.87 (39.15) | 1558.32 (64.95)
  Day 5 | 843.03 (12.00) | 1183.61 (51.92)

10. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to the Last Quantifiable Time Point After Single and Multiple Doses of Azacitidine
Description: The area under the plasma concentration-time curve from time zero to the last quantifiable time point (AUC0-t) of azacitidine following a single dose (Day 1) and multiple doses (Day 5) was calculated by the linear trapezoidal rule for participants with normal renal function and for participants with severe renal impairment.
Time Frame: Day 1 and Day 5: predose, 5, 15, 30, 45 minutes and 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, and 8 hours post-dose
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Normal RF: Azacitidine 75 mg/m^2 | Severe RI: Azacitidine 75 mg/m^2
Number analyzed (Participants) | 6 | 6
ng*hr/mL
  Day 1 | 920.76 (39.20) | 1558.72 (65.02)
  Day 5 | 841.62 (11.83) | 1181.83 (51.98)
Statistical Analysis 1: Comparison: Normal RF: Azacitidine 75 mg/m^2 vs Severe RI: Azacitidine 75 mg/m^2; Comparison of AUC0-t after a single dose (Day 1) in participants with normal renal function and participants with severe renal impairment. Geometric means, ratio and 90% CI of ratio of geometric means are from an analysis of variance model with renal function group (normal and severe), visit (Day 1 and Day 5), renal function group by visit interaction as fixed effect, and patient nested within renal function group as a random effect on the nature log-transformed pharmacokinetic parameters; Test type: Superiority or Other; Ratio (%) of Geometric Means = 169.3, 90% CI 2-sided [109.2 to 262.5] — Ratio of geometric mean is calculated as Severe RI/Normal RF and expressed as a percentage
Statistical Analysis 2: Comparison: Normal RF: Azacitidine 75 mg/m^2 vs Severe RI: Azacitidine 75 mg/m^2; Comparison of AUC0-t after multiple doses (Day 5) in participants with normal renal function and participants with severe renal impairment. Geometric means, ratio and 90% CI of ratio of geometric means are from an analysis of variance model with renal function group (normal and severe), visit (Day 1 and Day 5), renal function group by visit interaction as fixed effect, and patient nested within renal function group as a random effect on the nature log-transformed pharmacokinetic parameters; Test type: Superiority or Other; Ratio (%) of Geometric Means = 140.4, 90% CI 2-sided [90.6 to 217.7] — Ratio of geometric mean is calculated as Severe RI/Normal RF and expressed as a percentage

11. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity After Single and Multiple Doses of Azacitidine
Description: The area under the plasma concentration-time curve from time zero to infinity (AUC0-inf) for azacitidine, after a single dose (Day 1) and multiple doses (Day 5), calculated by the linear trapezoidal rule and extrapolated to infinity according to the following equation:
  AUC0-inf = AUC0-t + (Ct/ke), where Ct is the last quantifiable concentration and ke = elimination rate constant.
Time Frame: Day 1 and Day 5: predose, 5, 15, 30, 45 minutes and 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, and 8 hours post-dose
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Normal RF: Azacitidine 75 mg/m^2 | Severe RI: Azacitidine 75 mg/m^2
Number analyzed (Participants) | 6 | 6
ng*hr/mL
  Day 1 | 946.22 (39.05) | 1573.82 (63.46)
  Day 5 | 857.64 (9.94) | 1210.92 (49.07)
Statistical Analysis 1: Comparison: Normal RF: Azacitidine 75 mg/m^2 vs Severe RI: Azacitidine 75 mg/m^2; Comparison of AUC0-inf after a single dose (Day 1) in participants with normal renal function and participants with severe renal impairment. Geometric means, ratio and 90% CI of ratio of geometric means are from an analysis of variance model with renal function group (normal and severe), visit (Day 1 and Day 5), renal function group by visit interaction as fixed effect, and patient nested within renal function group as a random effect on the nature log-transformed pharmacokinetic parameters; Test type: Superiority or Other; Ratio (%) of Geometric Means = 166.3, 90% CI 2-sided [108.6 to 254.6] — Ratio of geometric mean is calculated as Severe RI/Normal RF and expressed as a percentage
Statistical Analysis 2: Comparison: Normal RF: Azacitidine 75 mg/m^2 vs Severe RI: Azacitidine 75 mg/m^2; Comparison of AUC0-inf after multiple doses (Day 5) in participants with normal renal function and participants with severe renal impairment. Geometric means, ratio and 90% CI of ratio of geometric means are from an analysis of variance model with renal function group (normal and severe), visit (Day 1 and Day 5), renal function group by visit interaction as fixed effect, and patient nested within renal function group as a random effect on the nature log-transformed pharmacokinetic parameters; Test type: Superiority or Other; Ratio (%) of Geometric Means = 141.2, 90% CI 2-sided [92.2 to 216.2] — Ratio of geometric mean is calculated as Severe RI/Normal RF and expressed as a percentage

12. Primary Outcome: Maximum Plasma Concentration of Azacitidine (Cmax) After Single and Multiple Doses of Azacitidine
Description: The maximum observed plasma concentration of azacitidine after a single dose (Day 1) or multiple doses (Day 5) for participants with normal renal function and for participants with severe renal impairment.
Time Frame: Day 1 and Day 5: predose, 5, 15, 30, 45 minutes and 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, and 8 hours post-dose
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Normal RF: Azacitidine 75 mg/m^2 | Severe RI: Azacitidine 75 mg/m^2
Number analyzed (Participants) | 6 | 6
ng/mL
  Day 1 | 745.50 (57.90) | 1056.66 (93.01)
  Day 5 | 632.56 (45.86) | 668.11 (91.64)
Statistical Analysis 1: Comparison: Normal RF: Azacitidine 75 mg/m^2 vs Severe RI: Azacitidine 75 mg/m^2; Comparison of Cmax after a single dose (Day 1) in participants with normal renal function and participants with severe renal impairment. Geometric means, ratio and 90% CI of ratio of geometric means are from an analysis of variance model with renal function group (normal and severe), visit (Day 1 and Day 5), renal function group by visit interaction as fixed effect, and patient nested within renal function group as a random effect on the nature log-transformed pharmacokinetic parameters; Test type: Superiority or Other; Ratio (%) of Geometric Means = 141.7, 90% CI 2-sided [73.2 to 274.6] — Ratio of geometric mean is calculated as Severe RI/Normal RF and expressed as a percentage
Statistical Analysis 2: Comparison: Normal RF: Azacitidine 75 mg/m^2 vs Severe RI: Azacitidine 75 mg/m^2; Comparison of Cmax after multiple doses (Day 5) in participants with normal renal function and participants with severe renal impairment. Geometric means, ratio and 90% CI of ratio of geometric means are from an analysis of variance model with renal function group (normal and severe), visit (Day 1 and Day 5), renal function group by visit interaction as fixed effect, and patient nested within renal function group as a random effect on the nature log-transformed pharmacokinetic parameters; Test type: Superiority or Other; Ratio (%) of Geometric Means = 105.6, 90% CI 2-sided [54.5 to 204.6] — Ratio of geometric mean is calculated as Severe RI/Normal RF and expressed as a percentage

13. Primary Outcome: Time to Maximum Plasma Concentration of Azacitidine (Tmax) After Single and Multiple Doses of Azacitidine
Description: The time to first maximum observed plasma concentration of azacitidine after a single dose (Day 1) or multiple doses (Day 5) for participants with normal renal function and severe renal impairment.
Time Frame: Day 1 and Day 5: predose, 5, 15, 30, 45 minutes and 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, and 8 hours post-dose
Population: as for outcome 9
Measure: Median (Full Range); unit: hours
Arm/Group | Normal RF: Azacitidine 75 mg/m^2 | Severe RI: Azacitidine 75 mg/m^2
Number analyzed (Participants) | 6 | 6
hours
  Day 1 | 0.25 [0.25 to 0.50] | 0.50 [0.25 to 1.50]
  Day 5 | 0.38 [0.25 to 0.50] | 0.64 [0.25 to 1.03]
Statistical Analysis 1: Comparison: Normal RF: Azacitidine 75 mg/m^2 vs Severe RI: Azacitidine 75 mg/m^2; Comparison of Tmax after a single dose (Day 1) in participants with normal renal function and participants with severe renal impairment; Test type: Superiority or Other; p = 0.1342, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.25, 90% CI 2-sided [0 to 0.52] — Median difference is Severe RI - Normal RF
Statistical Analysis 2: Comparison: Normal RF: Azacitidine 75 mg/m^2 vs Severe RI: Azacitidine 75 mg/m^2; Comparison of Tmax after multiple doses (Day 5) in participants with normal renal function and participants with severe renal impairment; Test type: Superiority or Other; p = 0.1017, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.25, 90% CI 2-sided [0 to 0.50] — Median difference is Severe RI - Normal RF

14. Primary Outcome: Terminal Phase Half-life of Azacitidine (t½) After Single and Multiple Doses of Azacitidine
Description: The terminal phase half-life of azacitidine after a single dose (Day 1) or multiple doses (Day 5) for participants with normal renal function and severe renal impairment, calculated according to the following equation: t½ = 0.693/λz, where λz is the terminal phase rate constant.
Time Frame: Day 1 and Day 5: predose, 5, 15, 30, 45 minutes and 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, and 8 hours post-dose
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Normal RF: Azacitidine 75 mg/m^2 | Severe RI: Azacitidine 75 mg/m^2
Number analyzed (Participants) | 6 | 6
hours
  Day 1 | 1.19 (102.56) [lower limit 102.56] | 0.97 (43.88)
  Day 5 | 1.03 (76.95) | 1.15 (53.86)

15. Primary Outcome: Apparent Total Clearance of Azacitidine (CL/F) After Single and Multiple Doses of Azacitidine
Description: The apparent total clearance of azacitidine after a single dose (Day 1) and multiple doses (Day 5) for participants with normal renal function and severe renal impairment, calculated as Dose/AUC0-inf.
Time Frame: Day 1 and Day 5: predose, 5, 15, 30, 45 minutes and 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, and 8 hours post-dose
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters/hour
Arm/Group | Normal RF: Azacitidine 75 mg/m^2 | Severe RI: Azacitidine 75 mg/m^2
Number analyzed (Participants) | 6 | 6
liters/hour
  Day 1 | 151.55 (30.88) | 85.76 (68.83)
  Day 5 | 166.95 (27.59) | 111.55 (51.75)

16. Primary Outcome: Apparent Volume of Distribution of Azacitidine (Vz/F) After Single and Multiple Doses of Azacitidine
Description: The apparent volume of distribution of azacitidine after a single dose (Day 1) and multiple doses (Day 5) for participants with normal renal function and severe renal impairment, calculated according to the equation: Vz/F = Apparent total clearance (CL/F) / terminal phase rate constant (λz).
Time Frame: Day 1 and Day 5: predose, 5, 15, 30, 45 minutes and 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, and 8 hours post-dose
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Normal RF: Azacitidine 75 mg/m^2 | Severe RI: Azacitidine 75 mg/m^2
Number analyzed (Participants) | 6 | 6
liters
  Day 1 | 259.44 (121.71) | 120.47 (120.45)
  Day 5 | 248.57 (115.10) | 184.54 (104.34)

17. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: A serious adverse event is one that at any dose of the study drug or at any time during the period of observation:
  * Results in death;
  * Is life threatening;
  * Requires inpatient hospitalization or prolongation of existing hospitalization;
  * Results in persistent or significant disability/incapacity;
  * Is a congenital anomaly/birth defect;
  * Is medically important.
  The Investigator assessed each AE for potential causal relationship between the event and study drug.
  The intensity of adverse changes in physical signs or symptoms was graded from 1 to 5 according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 3, and according to the following: Mild (Grade 1), Moderate (Grade 2), Severe (Grade 3), Life threatening (Grade 4), or Death (Grade 5).
Time Frame: Initial treatment phase: Days 1-11 for participants who received a single dose; Days 1-29 for participants who received multiple doses. Extension treatment period: From the date of first dose until 28 days after the date of last dose (up to 7 months).
Population: Safety population, all enrolled patients who received at least one dose of azacitidine and who had at least one post-treatment safety assessment.
Measure: Number; unit: participants
Arm/Group | Azacitidine 25 mg/m^2 | Azacitidine 50 mg/m^2 | Azacitidine 75 mg/m^2 | Azacitidine 100 mg/m^2 | Severe RI: Azacitidine 75 mg/m^2 | Extension Phase: Normal RF | Extension Phase: Severe RI
Number analyzed (Participants) | 5 | 5 | 6 | 5 | 6 | 14 | 4
participants
  Any adverse event | 4 | 3 | 6 | 5 | 6 | 14 | 4
  Adverse event related to study drug | 2 | 3 | 4 | 4 | 3 | 8 | 2
  Serious adverse event | 0 | 0 | 4 | 1 | 1 | 8 | 3
  Serious adverse event related to study drug | 0 | 0 | 0 | 1 | 0 | 1 | 1
  Grade 3 or 4 adverse event | 0 | 0 | 4 | 1 | 3 | 10 | 3
  AE leading to study drug discontinuation | 0 | 0 | 0 | 0 | 0 | 4 | 2
  AE leading to study drug interruption | 0 | 0 | 0 | 0 | 0 | 4 | 1
  AE leading to a dose reduction | 0 | 0 | 0 | 0 | 0 | 1 | 0
  AE leading to other action taken | 2 | 1 | 6 | 4 | 5 | 10 | 3
  Death | 0 | 0 | 0 | 0 | 0 | 1 | 1

ADVERSE EVENTS:
Time Frame: Initial treatment phase: Days 1-11 for participants who received a single dose; Days 1-29 for participants who received multiple doses. Extension treatment period: From the date of first dose until 28 days after the date of last dose (up to 7 months).
Arm/Group | Azacitidine 25 mg/m^2 | Azacitidine 50 mg/m^2 | Azacitidine 75 mg/m^2 | Azacitidine 100 mg/m^2 | Severe RI: Azacitidine 75 mg/m^2 | Extension Phase: Normal RF | Extension Phase: Severe RI
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 4/6 | 1/5 | 1/6 | 8/14 | 3/4
Other Adverse Events (participants affected / at risk) | 4/5 | 3/5 | 5/6 | 5/5 | 6/6 | 9/14 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Azacitidine 25 mg/m^2 (N=5) | Azacitidine 50 mg/m^2 (N=5) | Azacitidine 75 mg/m^2 (N=6) | Azacitidine 100 mg/m^2 (N=5) | Severe RI: Azacitidine 75 mg/m^2 (N=6) | Extension Phase: Normal RF (N=14) | Extension Phase: Severe RI (N=4)
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Renal vein thrombosis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Device dislocation (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Post procedural fistula (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Azacitidine 25 mg/m^2 (N=5) | Azacitidine 50 mg/m^2 (N=5) | Azacitidine 75 mg/m^2 (N=6) | Azacitidine 100 mg/m^2 (N=5) | Severe RI: Azacitidine 75 mg/m^2 (N=6) | Extension Phase: Normal RF (N=14) | Extension Phase: Severe RI (N=4)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 2 | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2 | 2 | 2
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 4 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 0 | 2 | 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Catheter site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Fatigue (General disorders) | 0 | 0 | 2 | 3 | 2 | 3 | 1
Gait disturbance (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hernia pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injection site discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Injection site erythema (General disorders) | 1 | 1 | 0 | 0 | 1 | 1 | 0
Injection site haematoma (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injection site haemorrhage (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Injection site induration (General disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0
Injection site pain (General disorders) | 0 | 2 | 1 | 1 | 2 | 0 | 0
Injection site pruritus (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Injection site rash (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Injection site reaction (General disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Injection site swelling (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Injection site vesicles (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Procedural site reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cardiac murmur (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Platelet count increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1 | 0 | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vaginal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Psychiatric symptom (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vulval disorder (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Peripheral coldness (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator shall have the right to publish and/or present study data provided that the investigator shall (i) furnish the sponsor a copy of any proposed publication or presentation generally thirty (30) days in advance of the submission, (ii) delete any confidential information of the sponsor, and (iii) delay submission for generally up to ninety (90) days to permit the preparation and filing of intellectual property applications or until sponsor gives its consent in a timely manner.